CLINICAL TRIAL: NCT06820762
Title: Irinotecan Liposome(II) Combined With Ivonescimab as Second-line Treatment for Small Cell Lung Cancer : A Prospective, Single-arm, Multicenter Clinical Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Shengjing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR070803-SCLC
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: SCLC
Keywords: SCLC，irinotecan liposome(II)，Ivonescimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Irinotecan liposome (II) combined with ivonescimab (Experimental): Subjects will be administered with irinotecan liposome(II) plus Ivonescimab via intravenously (IV) Q3W for 4-6 cycles, followed by Ivonescimab until disease progression or intolerable toxicity
  Interventions: Drug: irinotecan liposome(II) plus Ivonescimab via intravenously (IV) Q3W for 4-6 cycles, followed by Ivonescimab until disease progression or intolerable toxicity

INTERVENTIONS:
Drug: irinotecan liposome(II) plus Ivonescimab via intravenously (IV) Q3W for 4-6 cycles, followed by Ivonescimab until disease progression or intolerable toxicity — Drug: ivonescimab 20mg/kg, IV, D1, Q3W
  Other Names:
  AK112 Drug: irinotecan liposome(II) 70mg/m^2, IV, D1, Q3W

SUMMARY:
This study will evaluate the efficacy and safety of irinotecan liposome(II) in combination with Ivonescimab as second line treatment for SCLC.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multicenter clinical study assessing the efficacy and safety of irinotecan liposome(II) in combination with Ivonescimab as second line treatment for SCLC who failed first-line platinum-based chemotherapy with or without checkpoint inhibitors therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically or cytologically confirmed SCLC;
3. Advanced SCLC who failed first-line platinum-based chemotherapy with or without checkpoint inhibitors;
4. The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;
5. Life expectancy of ≥3 months;
6. At least one measurable lesion is present according to the efficacy evaluation criteria for RECIST 1.1（Lesions that have received radiotherapy within 6 months prior to the first dose cannot be used as target lesions）
7. No untreated central nervous system (CNS) metastases or CNS were stable for ≥1 month after treatment
8. Have adequate organ function;
9. All female must have had a negative serum pregnancy test within 72 hours of the first dosing and not be lactating, and study participants and their partners must use effective contraception during the trial and for 6 months after the last dosing of the trial drug.
10. Able and willing to provide a written informed consent;

Exclusion Criteria:

1. Known allergy to irinotecan hydrochloride liposome injection (II) and eboxizumab or drug excipients
2. History of severe active autoimmune disease
3. Participated in other drug studies within 4 weeks before enrollment
4. Imaging during the screening period showed that the tumor surrounded important blood vessels or had significant necrosis and voids, and the investigators determined that entering the study would cause bleeding risk
5. History of major illness within 1 year before the first medication
6. History of esophageal and gastric varices, severe ulcers, unhealed wounds, abdominal fistula, intraperitoneal abscess, or acute gastrointestinal bleeding within 6 months prior to initial administration
7. History of surgery or severe trauma within 4 weeks prior to initial dosing
8. Evidence and history of severe bleeding tendency;
9. Participants who had received or planned to receive a live vaccine within 4 weeks prior to the first study treatment
10. Patients with other cancer in 3 years,exceptions are adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
11. History of alcohol abuse, psychotropic substance abuse or drug abuse. Other conditions considered unsuitable for this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression or death due to any cause, whichever occurs first (based on RECIST v1.1).

SECONDARY OUTCOMES:
Objective response rate（ORR） | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.
Disease control rate (DCR) | Up to approximately 2 years
  DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks), based on RECIST v1.1.
Overall survival (OS) | Up to approximately 2 years
  OS is the time from the date of randomization or first dosing date to death due to any cause.
Treatment related adverse events (TRAEs) | Up to 30 days after last treatment
  The incidence and severity of TRAEs graded according to NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zheng, MD, Principal Investigator — Shengjing Hospital; Zhaoxia Dai, MD, Principal Investigator — The Second Affiliated Hospital of Dalian Medical University
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Spigel DR, Dowlati A, Chen Y, Navarro A, Yang JC, Stojanovic G, Jove M, Rich P, Andric ZG, Wu YL, Rudin CM, Chen H, Zhang L, Yeung S, Benzaghou F, Paz-Ares L, Bunn PA; RESILIENT Trial Investigators. RESILIENT Part 2: A Randomized, Open-Label Phase III Study of Liposomal Irinotecan Versus Topotecan in Adults With Relapsed Small Cell Lung Cancer. J Clin Oncol. 2024 Jul 1;42(19):2317-2326. doi: 10.1200/JCO.23.02110. Epub 2024 Apr 22. PMID 38648575
- [Background] Chen Z, Wu L, Wang Q, Yu Y, Liu X, Ma R, Li T, Li Y, Song X, Li L, Zhao W, Wang Q, Xu X, Lu S. Brief Report: Ivonescimab Combined With Etoposide Plus Carboplatin as First-Line Treatment for Extensive-Stage SCLC: Results of a Phase 1b Clinical Trial. J Thorac Oncol. 2025 Feb;20(2):233-239. doi: 10.1016/j.jtho.2024.10.013. Epub 2024 Oct 28. PMID 39490738
- [Background] Li L, Liu T, Liu Q, Mu S, Tao H, Yang X, Li Y, Xiong Q, Wang L, Hu Y. Rechallenge of immunotherapy beyond progression in patients with extensive-stage small-cell lung cancer. Front Pharmacol. 2022 Sep 6;13:967559. doi: 10.3389/fphar.2022.967559. eCollection 2022. PMID 36147357